CLINICAL TRIAL: NCT06780683
Title: Efficacy and Safety of Upadacitinib in the Treatment of Inflammatory Bowel Disease in China: a Multicenter, Single-Arm, Prospective, Observational Real-World Study
Brief Title: Efficacy and Safety of Upadacitinib in Inflammatory Bowel Disease
Acronym: EaseUpIBD
Status: Recruiting | Type: Observational
Sponsor: Xiang Gao (Other)
Responsible Party: Sponsor-Investigator, Xiang Gao, Director of Gastroenterology, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Other Study IDs: 2024ZSLYEC-250
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Fecal samples, serum samples, and tissue samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Crohn's disease
  Interventions: Drug: Upadacitinib
- ulcerative colitis
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Induction Therapy: The dose of upadacitinib for induction therapy is 45mg once daily for a duration of 8 weeks (for ulcerative colitis) or 12 weeks (for Crohn's disease).
  Maintenance Therapy: The dose of upadacitinib for maintenance therapy is 15mg once daily; for patients with refractory, severe, or extensive disease, a maintenance dose of 30mg once daily may be considered.

SUMMARY:
Inflammatory Bowel Disease (IBD), which encompasses ulcerative Colitis (UC) and Crohn's Disease (CD), has seen significant improvements in patient outcomes with biologic treatments. However, nearly half of the patients are either primary or secondary non-responders to the existing biologics. Upadacitinib is the only oral small molecule targeted drug approved for IBD in China. There is a paucity of research on the efficacy and safety of upadacitinib in treating Chinese patients with UC and CD, and a lack of study data on the Chinese IBD population. This study aims to conduct a multicenter, single-arm, prospective, observational real-world study to analyze the efficacy and safety of upadacitinib in the treatment of Chinese patients with IBD, providing a basis for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were patients of any gender, diagnosed with ulcerative colitis or Crohn's disease according to current guidelines, requiring initial upadacitinib treatment as judged by the treating physician, and providing signed informed consent.

Exclusion Criteria:

* Exclusion criteria included current or planned participation in any other clinical study, contraindications to upadacitinib treatment as per the drug's instructions, and patients deemed unsuitable for the study by the researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was derived from IBD centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission Rate | 52 weeks
  Clinical remission rate in patients with ulcerative Colitis or Crohn's Disease.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Ruikang Hospital Affiliated to Guangxi University of Chinese Medicine, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loftus EV Jr, Panes J, Lacerda AP, Peyrin-Biroulet L, D'Haens G, Panaccione R, Reinisch W, Louis E, Chen M, Nakase H, Begun J, Boland BS, Phillips C, Mohamed MF, Liu J, Geng Z, Feng T, Dubcenco E, Colombel JF. Upadacitinib Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2023 May 25;388(21):1966-1980. doi: 10.1056/NEJMoa2212728. PMID 37224198
- [Background] Danese S, Vermeire S, Zhou W, Pangan AL, Siffledeen J, Greenbloom S, Hebuterne X, D'Haens G, Nakase H, Panes J, Higgins PDR, Juillerat P, Lindsay JO, Loftus EV Jr, Sandborn WJ, Reinisch W, Chen MH, Sanchez Gonzalez Y, Huang B, Xie W, Liu J, Weinreich MA, Panaccione R. Upadacitinib as induction and maintenance therapy for moderately to severely active ulcerative colitis: results from three phase 3, multicentre, double-blind, randomised trials. Lancet. 2022 Jun 4;399(10341):2113-2128. doi: 10.1016/S0140-6736(22)00581-5. Epub 2022 May 26. PMID 35644166